CLINICAL TRIAL: NCT04662021
Title: The Effect of Aerobic Training Versus Cognitive Behavioral Therapy in Management of Anxiety, Depression and Stress-related to Covid 19 Pandemics Among University Students: a Comparative Study
Brief Title: Aerobic Training Versus Cognitive Behavioral Therapy in Management of Anxiety
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Marwa Eid, assistant professor of physical therapy for surgery, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 12-2020
Record Dates: First submitted 2020-12-04; First posted 2020-12-10 (Actual); Last update posted 2021-01-11 (Actual); Status verified 2021-01

CONDITIONS: Anxiety Depression Disorder
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise group (Experimental)
  Interventions: Other: Aerobic Exercises
- Cognitive therapy group (Experimental)
  Interventions: Other: Aerobic Exercises

INTERVENTIONS:
Other: Aerobic Exercises — Participants perform one hour of regular moderate to vigorous physical activities about (70 % to 90 %) of the maximum heart rate which was calculated according to this formula (HR max= 220- age)

SUMMARY:
Anxiety and depression disorders (ADD) have the highest overall prevalence rate among psychiatric disorders in young females. Its manifestations are disabling, distressing a substantial negative impact on the quality of life. The purpose of this study was to compare the effect of cognitive-behavioral therapy and physical therapy on female students with mild to moderate anxiety and depression.

DETAILED DESCRIPTION:
Female students of Taif University will be invited to participate in this study. 40 students will be assigned according to sample size calculation into the study as having mild to moderate anxiety and depression according to Depression, Anxiety and Stress Scale (DASS 21) most days of the week for at least six months. All study participants will sign an informed consent form. Screening for the physical activities in the last 7 days of all participants will be performed one day before starting the study protocol using The International Physical Activity Questionnaires (IPAQ) short form. The exclusion will be performed to severe psychological conditions such as schizophrenia and severe depression and any physical condition that limit physical activities. Also, participants who are taking any medications for the treatment of anxiety and depression will be excluded. Also, participants who had any abnormalities of the cardiovascular status that prevent them to perform the physical activities or reaching the target heart rate without risk as recommended by their primary care physician. The age range will be 18 to 25 years with a mean age of 21±0.75 years. Participants will be assigned into two groups: group A (GA) consists of 20 students and they will be instructed to increase their physical activities one hour daily, 5 days per week for 8 weeks of moderate to vigorous activities such as running, jumping, swimming, aerobics or dancing; and group B (GB) consists of 20 students and they will receive cognitive behavioral therapy for 8 sessions (once per week for 8 weeks).

ELIGIBILITY:
Inclusion Criteria:

* mild to moderate anxiety and depression according to Depression, Anxiety and Stress Scale (DASS 21) most days of the week for at least six months
* Females Age 18-25 years

Exclusion Criteria:

* severe psychological conditions such as schizophrenia
* severe depression
* any physical condition that limit physical activities

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2020-12-10 (Actual); Primary Completion 2021-02-10 (Estimated); Study Completion 2021-02-25 (Estimated)

PRIMARY OUTCOMES:
DASS 21 | 8 weeks
  The DASS 21 is a 21 item self-report questionnaire designed to measure the severity of a range of symptoms common to both Depression and Anxiety

CONTACTS AND LOCATIONS:
Locations (1):
- Marwa Eid, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No